CLINICAL TRIAL: NCT01323517
Title: A Phase II Trial of The Addition of Ipilimumab (MDX-010) To Isolated Limb Infusion (ILI) With Standard Melphalan and Dactinomycin In The Treatment of Advanced Unresectable Melanoma of The Extremity
Brief Title: Addition of Ipilimumab (MDX-010) To Isolated Limb Infusion (ILI) With Standard Melphalan and Dactinomycin In The Treatment of Advanced Unresectable Melanoma of The Extremity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-101
Record Dates: First submitted 2011-03-23; First posted 2011-03-25 (Estimated); Results first posted 2018-05-15 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2017-12

CONDITIONS: Melanoma
Keywords: skin; DACTINOMYCIN; MDX-010 (Ipilimumab); MELPHALAN; Isolated Limb Infusion; 10-101
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Melphalan; Dactinomycin

ARMS (1):
- Ipilimumab, Melphalan and Dactinomycin (Experimental): This is a single-institution phase II trial with a primary outcome of progression free survival (PFS).
  Interventions: Drug: Ipilimumab, Melphalan and Dactinomycin

INTERVENTIONS:
Drug: Ipilimumab, Melphalan and Dactinomycin — Isolated limb infusion ((ILI) with Melphalan and Dactinomycin- MSKCC operating room. Ipilimumab- IV administration in outpatient chemotherapy clinic. Induction therapy with Ipilimumab will start 1-3 weeks after ILI in the standard dose of 10mg/kg every 3 weeks for a total of 4 doses. Patients will then receive chronic therapy every 3 months. Patients will be followed every 3 months for 2 years.

SUMMARY:
The purpose of this study is to see the effect of adding a systemic study drug, Ipilimumab, to two standard chemotherapy drugs, Melphalan and Dactinomycin. The study drug Ipilimumab is an antibody to a normal protein found in the body, CTLA-4. This protein normally allows the immune system (the body's natural defense system that helps fight infections) uses to quiet an immune response. The study drug works by blocking this protein and allowing the immune system to become more active. This study will investigate the effects, of combining ILI (using two standard drugs to treat melanoma, Melphalan and Dactinomycin), with the study drug, Ipilimumab on advanced Melanoma cancer.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent.
* Histologic diagnosis of melanoma with in transit metastasis Stage IIIB, IIIC, or IV
* Required values for initial laboratory tests:
* WBC ≥ 2000/uL
* ANC ≥ 1000/uL
* Platelets ≥ 50 x 103/uL
* Hemoglobin ≥ 8 g/dL
* Creatinine ≤ 3.0 x ULN
* AST/ALT ≤ 2.5 x ULN
* Bilirubin ≤ 3.0 x ULN, (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
* No active or chronic infection with HIV, Hepatitis B, or Hepatitis C.
* Karnofsky performance status ≥60
* Men and women, ≥ 18 years of age. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal. Post-menopause is defined as:
* Amenorrhea ≥ 12 consecutive months without another cause, or
* For women with irregular menstrual periods and taking hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level ≥ 35 mIU/mL.
* Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of ipilimumab.

Exclusion Criteria:

* Any other malignancy form which the patient has been disease-free for less than 2 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix.
* Autoimmune disease: Patients with a history of inflammatory bowel disease are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome).
* Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
* Patients with underlying heart conditions who are deemed ineligible for surgery by cardiology consult
* Any history of prior treatment with ipilimumab or prior CD137 agonist or CTLA-4 inhibitor or agonist.
* Concomitant therapy with any of the following: IL-2, interferon, or other non-study immunotherapy regimens; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids.
* Women of childbearing potential (WOCBP), who:
* are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 8 weeks after cessation of study drug, or
* have a positive pregnancy test at baseline, or
* are pregnant or breastfeeding.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg, infectious) illness.
* Persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 8 weeks after ipilimumab is stopped.
* Sexually active WOCBP must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. Before study enrollment, WOCBP must be advised of the importance of avoiding pregnancy during study participation and the potential risk factors for an unintentional pregnancy. All WOCBP MUST have a negative pregnancy test before first receiving ipilimumab. If the pregnancy test is positive, the patient must not receive ipilimumab and must not be enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Ariyan, MD,PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ipilimumab, Melphalan and Dactinomycin
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ipilimumab, Melphalan and Dactinomycin
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 64 [37 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival at One Year.
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 1 year
Measure: Number; unit: percentage of participants PFS at 1 year
Arm/Group | Ipilimumab, Melphalan and Dactinomycin
Number analyzed (Participants) | 26
percentage of participants PFS at 1 year | 58

2. Secondary Outcome: Toxicity of Additional Ipilimumab Will be Evaluated for All Treated Patients Using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab, Melphalan and Dactinomycin
Number analyzed (Participants) | 26
Participants | 26

3. Secondary Outcome: To Determine Response Rates of Combination Therapy. Tumor Assessment Will be Measured by the Immune Related Response Criteria (irRC).
Description: Progression free survival, from time of ILI, will be determined by measuring the index lesions, non-index lesions, and new lesions as described below. Patients with deep lesions will have repeat CT Scan evaluation to quantitate the lesions.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab, Melphalan and Dactinomycin
Number analyzed (Participants) | 24
Participants
  Complete Response | 16
  Partial Response | 5
  Stable Disease | 1
  Progressive Disease | 2

4. Secondary Outcome: To Define the Immunologic Events and Signatures at the Tumor Site and in the Periphery That Corresponds to Response to Ipilimumab.
Description: Summaries of antibody response, comparison of pretreatment with post-ipilimumab and end of treatment will be assessed for percent of CD4, CD8, and CD68 positive cells
Time Frame: 2 years
Measure: Mean (Full Range); unit: percent of positive cells
Arm/Group | Ipilimumab, Melphalan and Dactinomycin
Number analyzed (Participants) | 26
percent of positive cells
  Pretreatment CD4 | 3 [1 to 17]
  Posttreatment CD4 | 28 [2 to 49]
  Pretreatment CD8 | 2 [1 to 5]
  Posttreatment CD8 | 7 [1 to 26]
  Pretreatment CD68 | 10 [1 to 19]
  Posttreatment CD68 | 18 [2 to 38]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Ipilimumab, Melphalan and Dactinomycin
All-Cause Mortality (participants affected / at risk) | 6/26
Serious Adverse Events (participants affected / at risk) | 10/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab, Melphalan and Dactinomycin (N=26)
Acute coronary syndrome (Cardiac disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Hypotension (Vascular disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Malaise (General disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Resp, thoracic & mediastinal disorder Other, spec (Respiratory, thoracic and mediastinal disorders) | 1
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 2
Sepsis (Infections and infestations) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Thromboembolic event (Vascular disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab, Melphalan and Dactinomycin (N=26)
Hyperglycemia (Metabolism and nutrition disorders) | 15
Hypocalcemia (Metabolism and nutrition disorders) | 12
Diarrhea (Gastrointestinal disorders) | 11
CPK increased (Investigations) | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 7
Papulopustular rash (Infections and infestations) | 6
Adrenal insufficiency (Endocrine disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Alanine aminotransferase increased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 4
Fatigue (General disorders) | 4
Hypothyroidism (Endocrine disorders) | 4
Aspartate aminotransferase increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Blood bilirubin increased (Investigations) | 3
Hyponatremia (Metabolism and nutrition disorders) | 3
Sinusitis (Infections and infestations) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Colitis (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Pain (General disorders) | 2
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Endocrine disorders - Other, specify (Endocrine disorders) | 2
Urinary tract infection (Infections and infestations) | 2
Stomach pain (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT01323517/Prot_SAP_000.pdf